CLINICAL TRIAL: NCT01826591
Title: Do Insulin Secretion or Genotype Pattern Predict Low Fat vs Low Carb Weight Loss Success?
Brief Title: DIETFITS Study (Diet Intervention Examining the Factors Interacting With Treatment Success
Acronym: DIETFITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Nutrition Science Initiative (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22305; 1R01DK091831 (NIH); T32HL007034 (NIH); UL1TR001085 (NIH)
Record Dates: First submitted 2013-03-27; First posted 2013-04-08 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Low-Carbohydrate Diet (Experimental): Healthy, Low-Carbohydrate Diet
  Interventions: Behavioral: Low-Carbohydrate Diet; Behavioral: Mobile App
- Experimental: Low-Fat Diet (Experimental): Healthy, Low-Fat Diet
  Interventions: Behavioral: Low-Fat Diet; Behavioral: Mobile App

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diet — Counseling/instruction on how to follow a low-carbohydrate diet.
  Arms: Experimental: Low-Carbohydrate Diet
Behavioral: Low-Fat Diet — Counseling/instruction on how to follow a low-fat diet.
  Arms: Experimental: Low-Fat Diet
Behavioral: Mobile App — Mobile app to increase vegetable consumption. Participants with iPhones will be re-randomized to receive a mobile app beginning at either months 4-5 or months 7-8. The first phase during months 4-7 will be used to compare the effect of a mobile app (intervention) vs. no mobile app (waiting-list control). The a priori hypothesis is that vegetable consumption will increase among those who receive the app in both diet groups.

SUMMARY:
Genomics research is advancing rapidly, and links between genes and obesity continue to be discovered and better defined. A growing number of single nucleotide polymorphisms (SNPs) in multiple genes have been shown to alter an individual's response to dietary macronutrient composition. Based on prior genetic studies evaluating the body's physiological responses to dietary carbohydrates or fats, the investigators identified multi-locus genotype patterns with SNPs from three genes (FABP2, PPARG, and ADRB2): a low carbohydrate-responsive genotype (LCG) and a low fat-responsive genotype (LFG). In a preliminary, retrospective study (using the A TO Z weight loss study data), the investigators observed a 3-fold difference in 12-month weight loss for initially overweight women who were determined to have been appropriately matched vs. mismatched to a low carbohydrate (Low Carb) or low fat (Low Fat) diet based on their multi-locus genotype pattern. The primary objective of this study is to confirm and expand on the preliminary results and determine if weight loss success can be increased if the dietary approach (Low Carb vs. Low Fat) is appropriately matched to an individual' s genetic predisposition (Low Carb Genotype vs. Low Fat Genotype) toward those diets.

DETAILED DESCRIPTION:
If the intriguing preliminary retrospective results are confirmed in this full scale study, the results will demonstrate that inexpensive DNA testing could help dieters predict whether they will have greater weight loss success on a Low Carb or a Low Fat diet. Commensurate with increasing scientific interest in personalized medicine approaches to intervention development, this would provide an example of the potentially substantial health impacts that could be obtained through understanding specific gene-environment interactions that have been anticipated from the unraveling of the human genome.

Mobile App Sub-Study-For the purpose of augmenting adherence to high vegetable consumption in both diet groups, we will develop a theory-based mobile app to increase vegetable consumption through goal-setting, self-monitoring, and social comparison. Participants from both diet groups with iPhones will be re-randomized to receive the app at either months 4-5 or months 7-8. The first phase during months 4-7 will be used to compare the effect of a mobile app (intervention) vs. no mobile app (waiting-list control). The a priori hypothesis is that vegetable consumption will increase among those who receive the app in both diet arms. The investigator and outcomes assessor will be blinded to group assignment. Intention-to-treat analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years of age
* Women: Pre-menopausal (self-report) and <50 years of age
* Men: <50 years of age
* BMI (body mass index): 27-40 kg/m2 (need to lose >10% body weight to achieve healthy BMI)
* Body weight stable for the last two months, and not actively on a weight loss plan
* No plans to move from the area over the next two years
* Available and able to participate in the evaluations and intervention for the study period
* Willing to accept random assignment
* To enhance study generalizability, people on medications not noted below as specific exclusions can
* participate if they have been stable on such medications for at least three months
* Ability and willingness to give written informed
* No known active psychiatric illness

Exclusion Criteria:

Subjects with the following conditions will be excluded (determined by self-report):

* Pregnant, lactating, within 6 months post-partum, or planning to become pregnant in the next 2 years
* Diabetes (type 1 and 2) or history of gestational diabetes or on hypoglycemic medications for any other indication
* Prevalent diseases: Malabsorption, renal or liver disease, active neoplasms, recent myocardial infarction (<6 months)(patient self-report and, if available, review of labs from primary care provider)
* Smokers (because of effect on weight and lipids)
* History of serious arrhythmias, or cerebrovascular disease
* Uncontrolled hyper- or hypothyroidism (TSH not within normal limits)
* Medications: Lipid lowering, antihypertensive medications, and those known to affect weight/energy expenditure
* Excessive alcohol intake (self-reported, >3 drinks/day)
* Musculoskeletal disorders precluding regular physical activity
* Unable to follow either of the two study diets for reasons of food allergies or other (e.g., vegan)
* Currently under psychiatric care, or taking psychiatric medications
* Inability to communicate effectively with study personnel

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 609 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight at 12 months | Baseline and 12 months
  Weight change was calculated as the 12 month value minus the baseline value. The study was designed to determine if either insulin secretion or genotype pattern (low-fat genotype pattern vs .low-carb genotype pattern) were significant effect modifiers of 12-month weight loss for the two diet arms (e.g., 2X2 analyses).

SECONDARY OUTCOMES:
Change from baseline in LDL cholesterol at 12 months | Baseline and 12 months
  LDL-cholesterol change was calculated as the 12 month value minus the baseline value.
Change from baseline in HDL cholesterol at 12 months | Baseline and 12 months
  HDL-cholesterol change was calculated as the 12 month value minus the baseline value.
Change from baseline in triglycerides at 12 months | Baseline and 12 months
  Triglycerides change was calculated as the 12 month value minus the baseline value.
Change from baseline in fasting insulin at 12 months | Baseline and 12 months
  Fasting insulin change was calculated as the 12 month value minus the baseline value.
Change from baseline in fasting glucose at 12 months | Baseline and 12 months
  Fasting glucose change was calculated as the 12 month value minus the baseline value.
Change from baseline in insulin after an oral-glucose tolerance test (OGTT) at 12 months | Baseline and 12 months
  Post-OGTT insulin change was calculated as the 12 month value minus the baseline value.
Change from baseline in glucose after an oral-glucose tolerance test (OGTT) at 12 months | Baseline and 12 months
  Post-OGTT glucose change was calculated as the 12 month value minus the baseline value.
Change from baseline in body fat percentage at 12 months. | Baseline and 12 months
  Body fat percentage was assessed by dual-energy x-ray absorptiometry (DXA) and the change was calculated as the 12 month value minus the baseline value.
Change from baseline in body mass index (BMI) at 12 months. | Baseline and 12 months
  BMI change was calculated as the 12 month value minus the baseline value.
Change from baseline in resting energy expenditure (REE) at 12 months. | Baseline and 12 months
  REE was assessed by indirect calorimetry and the change was calculated as the 12 month value minus the baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mummah SA, Robinson TN, King AC, Gardner CD, Sutton S. IDEAS (Integrate, Design, Assess, and Share): A Framework and Toolkit of Strategies for the Development of More Effective Digital Interventions to Change Health Behavior. J Med Internet Res. 2016 Dec 16;18(12):e317. doi: 10.2196/jmir.5927. PMID 27986647
- [Background] Mummah SA, Mathur M, King AC, Gardner CD, Sutton S. Mobile Technology for Vegetable Consumption: A Randomized Controlled Pilot Study in Overweight Adults. JMIR Mhealth Uhealth. 2016 May 18;4(2):e51. doi: 10.2196/mhealth.5146. PMID 27193036
- [Background] Mummah SA, King AC, Gardner CD, Sutton S. Iterative development of Vegethon: a theory-based mobile app intervention to increase vegetable consumption. Int J Behav Nutr Phys Act. 2016 Aug 8;13:90. doi: 10.1186/s12966-016-0400-z. PMID 27501724
- [Background] Stanton MV, Robinson JL, Kirkpatrick SM, Farzinkhou S, Avery EC, Rigdon J, Offringa LC, Trepanowski JF, Hauser ME, Hartle JC, Cherin RJ, King AC, Ioannidis JP, Desai M, Gardner CD. DIETFITS study (diet intervention examining the factors interacting with treatment success) - Study design and methods. Contemp Clin Trials. 2017 Feb;53:151-161. doi: 10.1016/j.cct.2016.12.021. Epub 2016 Dec 24. PMID 28027950
- [Background] Gardner CD, Trepanowski JF, Del Gobbo LC, Hauser ME, Rigdon J, Ioannidis JPA, Desai M, King AC. Effect of Low-Fat vs Low-Carbohydrate Diet on 12-Month Weight Loss in Overweight Adults and the Association With Genotype Pattern or Insulin Secretion: The DIETFITS Randomized Clinical Trial. JAMA. 2018 Feb 20;319(7):667-679. doi: 10.1001/jama.2018.0245. PMID 29466592
- [Background] Shih CW, Hauser ME, Aronica L, Rigdon J, Gardner CD. Changes in blood lipid concentrations associated with changes in intake of dietary saturated fat in the context of a healthy low-carbohydrate weight-loss diet: a secondary analysis of the Diet Intervention Examining The Factors Interacting with Treatment Success (DIETFITS) trial. Am J Clin Nutr. 2019 Feb 1;109(2):433-441. doi: 10.1093/ajcn/nqy305. PMID 30649213
- [Background] Fielding-Singh P, Patel ML, King AC, Gardner CD. Baseline Psychosocial and Demographic Factors Associated with Study Attrition and 12-Month Weight Gain in the DIETFITS Trial. Obesity (Silver Spring). 2019 Dec;27(12):1997-2004. doi: 10.1002/oby.22650. Epub 2019 Oct 21. PMID 31633313
- [Background] Grembi JA, Nguyen LH, Haggerty TD, Gardner CD, Holmes SP, Parsonnet J. Gut microbiota plasticity is correlated with sustained weight loss on a low-carb or low-fat dietary intervention. Sci Rep. 2020 Jan 29;10(1):1405. doi: 10.1038/s41598-020-58000-y. PMID 31996717
- [Background] Figarska SM, Rigdon J, Ganna A, Elmstahl S, Lind L, Gardner CD, Ingelsson E. Proteomic profiles before and during weight loss: Results from randomized trial of dietary intervention. Sci Rep. 2020 May 13;10(1):7913. doi: 10.1038/s41598-020-64636-7. PMID 32404980
- [Derived] Lai CQ, Parnell LD, Das SK, Gardner CD, Ordovas JM. Differential weight-loss responses of APOA2 genotype carriers to low-carbohydrate and low-fat diets: the DIETFITS trial. Obesity (Silver Spring). 2025 Jun;33(6):1048-1057. doi: 10.1002/oby.24288. Epub 2025 May 1. PMID 40310284
- [Derived] Krauss RM, Fisher LM, King SM, Gardner CD. Changes in soluble LDL receptor and lipoprotein fractions in response to diet in the DIETFITS weight loss study. J Lipid Res. 2024 Mar;65(3):100503. doi: 10.1016/j.jlr.2024.100503. Epub 2024 Jan 19. PMID 38246235
- [Derived] Hauser ME, Hartle JC, Landry MJ, Fielding-Singh P, Shih CW, Qin F, Rigdon J, Gardner CD. Association of dietary adherence and dietary quality with weight loss success among those following low-carbohydrate and low-fat diets: a secondary analysis of the DIETFITS randomized clinical trial. Am J Clin Nutr. 2024 Jan;119(1):174-184. doi: 10.1016/j.ajcnut.2023.10.028. Epub 2023 Nov 4. PMID 37931749
- [Derived] Soto-Mota A, Pereira MA, Ebbeling CB, Aronica L, Ludwig DS. Evidence for the carbohydrate-insulin model in a reanalysis of the Diet Intervention Examining The Factors Interacting with Treatment Success (DIETFITS) trial. Am J Clin Nutr. 2023 Mar;117(3):599-606. doi: 10.1016/j.ajcnut.2022.12.014. Epub 2023 Jan 6. PMID 36811468
- [Derived] Hartle JC, Zawadzki RS, Rigdon J, Lam J, Gardner CD. Development and evaluation of a novel dietary bisphenol A (BPA) exposure risk tool. BMC Nutr. 2022 Dec 6;8(1):143. doi: 10.1186/s40795-022-00634-4. PMID 36474269
- [Derived] Cauwenberghs N, Prunicki M, Sabovcik F, Perelman D, Contrepois K, Li X, Snyder MP, Nadeau KC, Kuznetsova T, Haddad F, Gardner CD. Temporal changes in soluble angiotensin-converting enzyme 2 associated with metabolic health, body composition, and proteome dynamics during a weight loss diet intervention: a randomized trial with implications for the COVID-19 pandemic. Am J Clin Nutr. 2021 Nov 8;114(5):1655-1665. doi: 10.1093/ajcn/nqab243. PMID 34375388
- [Derived] Fragiadakis GK, Wastyk HC, Robinson JL, Sonnenburg ED, Sonnenburg JL, Gardner CD. Long-term dietary intervention reveals resilience of the gut microbiota despite changes in diet and weight. Am J Clin Nutr. 2020 Jun 1;111(6):1127-1136. doi: 10.1093/ajcn/nqaa046. PMID 32186326
- [Derived] Oppezzo MA, Stanton MV, Garcia A, Rigdon J, Berman JR, Gardner CD. To Text or Not to Text: Electronic Message Intervention to Improve Treatment Adherence Versus Matched Historical Controls. JMIR Mhealth Uhealth. 2019 Apr 9;7(4):e11720. doi: 10.2196/11720. PMID 30964436
- [Derived] Guo J, Robinson JL, Gardner CD, Hall KD. Objective versus Self-Reported Energy Intake Changes During Low-Carbohydrate and Low-Fat Diets. Obesity (Silver Spring). 2019 Mar;27(3):420-426. doi: 10.1002/oby.22389. Epub 2019 Jan 22. PMID 30672127
- [Derived] Mummah S, Robinson TN, Mathur M, Farzinkhou S, Sutton S, Gardner CD. Effect of a mobile app intervention on vegetable consumption in overweight adults: a randomized controlled trial. Int J Behav Nutr Phys Act. 2017 Sep 15;14(1):125. doi: 10.1186/s12966-017-0563-2. PMID 28915825
- See also: Study description and results summary — https://med.stanford.edu/nutrition/research/completed-studies/diet-study.html